CLINICAL TRIAL: NCT02851927
Title: Rigid 'Mini-thoracoscopy' vs Semirigid Thoracoscopy in Undiagnosed Exudative Pleural Effusions : A Randomized Controlled Trial
Brief Title: Mini Thoracoscopy vs Semirigid Thoracoscopy in Exudative Pleural Effusions
Acronym: MIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Karan Madan, Dr Karan Madan MD, DM Assistant Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Mini vs Semirigid RCT
Record Dates: First submitted 2016-05-01; First posted 2016-08-02 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mini Thoracoscopy (Experimental): Thoracoscopy procedure shall be performed using the Rigid Mini Thoracoscope
  Interventions: Procedure: Mini Thoracoscopy
- Semirigid Thoracoscopy (Active Comparator): Thoracoscopy procedure shall be performed using the SemiRigid Thoracoscope
  Interventions: Procedure: SemiRigid Thoracoscopy

INTERVENTIONS:
Procedure: Mini Thoracoscopy — Pleural biopsy using rigid mini thoracoscope
  Arms: Mini Thoracoscopy
Procedure: SemiRigid Thoracoscopy — Pleural biopsy using semirigid thoracoscope
  Arms: Semirigid Thoracoscopy

SUMMARY:
Undiagnosed pleural effusion is a diagnostic dilemma especially in exudative pleural effusions (EPE). 20-40 % are unable to be attributed to a specific diagnosis, even after thoracentesis and closed pleural biopsy. Thoracoscopy has been demonstrated to increase the diagnostic yield in undiagnosed EPE. The diagnostic yield of thoracoscopy in malignant and TB pleural effusion ranges from 91% to 94% and 93% to 100%, respectively.

Rigid thoracoscopy has traditionally been the modality of choice. The recently introduced semirigid thoracoscope provides ease of handling like a flexible bronchoscope. However, there are concerns about the diagnostic yield of semi-rigid thoracoscopy when compared with rigid thoracoscopy. According to the available literature, the yield of semirigid and rigid thoracoscopy is almost similar if adequate pleural biopsy is obtained. However there are concerns that with semi-rigid thoracoscope, there might be greater incidence of inability to obtain adequate pleural biopsy. On the other hand, the use of conventional rigid thoracoscope may be associated with greater procedure related pain.Mini-Thoracoscopy is a newer rigid thoracoscopy instrument which is smaller in diameter (5.5 mm) and may allow pleural biopsy with a smaller incision. There is scant literature on its utility. The investigators hereby propose to undertake a randomized comparison of rigid 'mini thoracoscope' vs semi rigid thoracoscope in undiagnosed pleural effusions.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria and giving prior consent for the study shall be randomised. The randomization sequence will be computer generated with variable block size and the assignments will be placed in opaque sealed envelopes. All patients will undergo hemogram, liver and renal function tests, coagulation profile, an electrocardiogram and Computed tomography (CT) of the chest before entering the study. Chest ultrasound will be performed in all patients to evaluate the rib spaces, amount of pleural fluid and for selection of the entry point.

Instruments The semi-rigid thoracoscope to be used is the autoclavable Olympus LTF-160 (Olympus, Tokyo, Japan) thoracoscope with 2.8 mm inner channel diameter and 7 mm outer diameter. The forceps is flexible forceps with alligator jaw with spike cusps, 2.8 mm of the outer diameter. The rigid mini thoracoscope is the Richard Wolf 5.5 mm operating endoscope with the working channel.

Thoracoscopy technique Thoracoscopy will be performed in the interventional pulmonology lab. Patients shall be fasting for solids for 8 hours and for liquids 6 hours. Patients shall be having continuous monitoring of blood pressure, pulse rate, and oxygen saturation.

Topical anesthesia will be achieved by infiltrating 2% lidocaine locally at the incision site. The procedure shall be performed under conscious sedation and analgesia using a combination of midazolam and intravenous fentanyl. An incision shall be made at the site of maximum fluid thickness as assessed by pre-procedural USG chest, with the patient in lateral decubitus position and involved side upward. After incision, the appropriately sized trocar shall be placed through the skin into the pleural space. The thoracoscope shall be inserted through the trocar. The pleural surfaces shall then be thoroughly inspected. A minimum of 6-8 pleural biopsy samples shall be obtained by semi-rigid thoracoscope and at least 4 with rigid mini-thoracoscope.

Samples shall be sent for histopathological analysis and mycobacterial cultures. At the end of the procedure, a chest tube shall be placed and removed subsequently.

All patients shall be followed up for a period of six months from the time of procedure if non-specific inflammation/ fibrinous pleuritis is the diagnosis or no definitive diagnosis is made during that time.

Statistical analysis:

Data shall be expressed as mean ± standard deviation (SD), or percentage. Differences in continuous variables between the two groups shall be compared using Student's t test (or Mann-Whitney U test); while differences in categorical data shall be compared using the chi-square test (or Fisher's exact test). A p value of less than 0.05 shall be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years Presence of undiagnosed exudative pleural effusion as determined by the criteria detailed by Light et al where a specific diagnosis was not obtained after initial cytological and/or microbiological examinations.

Adequate rib spaces for successful performance of thoracoscopy as judged by clinical examination Adequate pleural fluid space as judged by pre-procedural USG chest

Exclusion Criteria:

1. Pregnancy
2. Coagulopathy (platelet count < 50000/mm3, INR > 1.5)
3. Unstable hemodynamic status ( SBP > 180, DBP> 100 or SBP< 90 mm Hg / heart failure
4. Myocardial infarction or unstable angina in the last 6 wk
5. Hypoxemia not correctable with low flow oxygen (SpO2 <90% despite low flow oxygen @ 1-2 l/min)
6. Extensive rib crowding as judged by clinical examination
7. Extensive adhesions and lack of pleural space on USG chest
8. Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield | Through study completion, an average of 1 year
  Proportion of diagnostic biopsies in the two arms

SECONDARY OUTCOMES:
Sedation dose | Through study completion, an average of 1 year
  Comparison of sedative and analgesic agent doses between the two groups
Complications | Through study completion, an average of 1 year
  Complications related to the procedure
Procedural pain | Through study completion, an average of 1 year
  Patient rated procedural pain on Visual Analogue Scale
Operator rated pain | Through study completion, an average of 1 year
  Operator rated procedural pain on Visual Analogue Scale
Operator rated overall procedure satisfaction | Through study completion, an average of 1 year
  Operator rated overall procedure satisfaction on Visual Analogue Scale
Biopsy Size | Through study completion, an average of 1 year
  Mean size of biopsy obtained during pleural biopsy procedure
Alternate equipment | Through study completion, an average of 1 year
  Requirement of conversion to alternate equipment for pleural biopsy
Image quality | Through study completion, an average of 1 year
  Operator rated image quality of pleural visualization (VAS)

OTHER OUTCOMES:
Ease of biopsy | Through study completion, an average of 1 year
  Ease of obtaining pleural biopsy on visual analogue scale
Operator rated pain on scope manipulation | Through study completion, an average of 1 year
  Operator rated pain on scope manipulation on Visual analogue scale (VAS)
Expectation of diagnostic biopsy | Through study completion, an average of 1 year
  Expectation that biopsy will be diagnostic on Visual Analogue Scale
Ease of manoeuvring thoracoscope | Through study completion, an average of 1 year
  Ease of scope maneuvering on Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Guleria, MD, DM, Study Chair — AIIMS, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided